CLINICAL TRIAL: NCT00908232
Title: Efficacy and Safety of Velcade Plus Dexamethasone (VD), VD+Cyclophosphamide or VD Plus Lenalidomide in MMY Patients Who Are Refractory or Have Relapsed After Their Primary Therapy for MMY and Have Achieved Stable Disease After 4 Cycles of VD
Brief Title: Treatment With Velcade (Bortezomib) Plus Dexamethasone (VD) or VD Plus Cyclophosphamide or VD Plus Lenalidomide in Patients With Multiple Myeloma Stabilized After 4 Cycles of VD
Acronym: SEQUENTIAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR013165; 26866138MMY2045 (Other: Janssen); 2007-001462-33 (EudraCT Number)
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Results first posted 2012-06-08 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; bortezomib; hematology; bone marrow cancer; immunoglobulin; refractory; progression; dexamethasone; lenalidomide; cyclophosphamide
MeSH Terms: conditions — Multiple Myeloma; Bone Marrow Neoplasms; Disease Progression | interventions — Cyclophosphamide; Bortezomib; Dexamethasone; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Stable Disease: VD (Experimental): Stable disease after 4 cycles bortezomib + dexamethasone: bortezomib 1.3 mg/m2 IV bolus on Day 1, 4, 8, 11 in combination with dexamethasone 20 mg orally daily, on Days 1, 2, 4, 5, 8, 9, 11, 12 for cycle 1 to 8
  Interventions: Drug: Bortezomib; Drug: Dexamethasone
- Stable Disease: VDC (Experimental): Stable disease after 4 cycles bortezomib + dexamethasone: bortezomib 1.3 mg/m2 IV bolus on Day 1, 4, 8 and 11 in combination with dexamethasone 20 mg orally daily, on Days 1, 2, 4, 5, 8, 9, 11, 12 for cycle 1 to 8 and cyclophosphamide 500 mg, orally daily, days 1, 8 and 15 for cycle 5 to 8
  Interventions: Drug: Cyclophosphamide; Drug: Bortezomib; Drug: Dexamethasone
- Stable Disease: VDL (Experimental): Stable disease after 4 cycles bortezomib + dexamethasone: bortezomib 1.3 mg/m2 IV bolus on Day 1, 4, 8 and 11 in combination with dexamethasone 20 mg orally daily, on Days 1, 2, 4, 5, 8, 9, 11, 12 for cycle 1 to 8 and lenalidomide 10 mg orally daily from day 1 to day 14 for cycle 5 to 8
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Lenalidomide
- Complete to Partial Response: VD (Experimental): Complete, very good partial or partial response after 4 cycles bortezomib + dexamethasone: bortezomib 1.3 mg/m2 IV bolus on Day 1, 4, 8, 11 in combination with dexamethasone 20 mg orally daily, on Days 1, 2, 4, 5, 8, 9, 11, 12 for cycle 1 to 8
  Interventions: Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Cyclophosphamide — 500 mg, p.o daily, days 1, 8 and 15 for cycles 5 to 8 cycles
  Arms: Stable Disease: VDC
Drug: Bortezomib — 1.3 mg/m2 IV bolus on Day 1, 4, 8, 11 for cycles 1 to 8
Drug: Dexamethasone — 20 mg orally daily, on Days 1, 2, 4, 5, 8, 9, 11, 12 for cycles 1 to 8
Drug: Lenalidomide — 10 mg orally daily, days 1-14 for cycles 5 to 8
  Arms: Stable Disease: VDL

SUMMARY:
The purpose of this study is to test the effectiveness and safety of adding cyclophosphamide or lenalidomide to the VD combination in the treatment of patients with multiple myeloma that have achieved a stable response after 4 initial cycles of treatment with VD. Multiple myeloma is the second most common cancer of the blood. Bortezomib disrupts the life cycle of the cell, affecting numerous biologic pathways, including those related to growth and survival of cancer cells.

DETAILED DESCRIPTION:
It has been shown that quality of response corresponds with clinical benefit. Stable disease is not regarded as a satisfactory result of therapy for relapsed and refractory multiple myeloma. However, there is no consensus if, when and how treatment should be continued or changed in the case of stable disease.

There are different strategies of achieving an optimal quality of response in relapsed and refractory multiple myeloma. One is to treat for a longer duration with one regimen. The alternative path can be a sequential approach adding another agent to the initial regimen depending on the outcome of therapy after a defined treatment period. These two principles will be evaluated in the present study.

Both Cyclophosphamide and Lenalidomide have proven to be efficacious in multiple myeloma and combinations of both agents with bortezomib and Dexamethasone have been shown to be active and tolerable.

In this study patients with relapsed/progressive or refractory multiple myeloma will start treatment with bortezomiib and Dexamethasone. Response will be evaluated after four cycles. Patients with complete, very good partial response or partial response will continue treatment as initiated. Patients with stable disease will either continue treatment with the bortezomib/Dexamethasone combination for another four cycles or will receive Cyclophosphamide or Lenalidomide as an additional third agent for another four cycles.

Patients with multiple myeloma that are refractory to or have relapsed/progressed after primary treatment for multiple myeloma will be enrolled in the study. All patients will receive a combination of bortezomib plus dexamethasone for a total of four cycles. Based on the response to this treatment, further study treatment is customized. Patients with a complete, a very good partial or a partial response will continue to receive bortezomib and Dexamethasone for a maximum additional four cycles, to an overall maximum of eight cycles. Patients achieving stable disease, as defined by International Myeloma Working Group 2006 (IMWG 2006) response criteria, will undergo a central randomisation to continue treatment with VD or VD plus cyclophosphamide or VD plus lenalidomide. Patients with progressive disease will go off study treatment. After randomisation, patients will receive therapy for up to four additional treatment cycles, to an overall maximum of eight cycles. Each cycle will consist of three weeks treatment. There will be a long-term follow-up period with monthly visits until relapse or progressive disease. Thereafter follow-up for survival will be continued by at least a phone call every other month. This will be performed for all patients until the last patient was treated and followed up for 1 year.

Safety will be assessed by the monitoring of adverse events, physical examination (including neurological/peripheral neurological examinations), pulmonary examinations, vital signs measurements, and clinical laboratory tests.

Patients will be treated in a 3-week cycle, up to a maximum of 8 cycles bortezomib 1.3 mg/m2 will be administered on day 1, 4, 8 and 11 as i.v. bolus infusion.

Dexamethasone 20 mg po will be administered on days 1, 2, 4, 5, 8, 9, 11, 12. Dexamethasone will be administered as 2 tables of 8 mg plus 1 tablet of 4 mg Cyclophosphamide 500 mg po will be administered as 10 tablets of 50 mg on day 1, 8, 15 Lenalidomide will be administered as once daily 10 mg tablet from day 1 to 14

ELIGIBILITY:
Inclusion Criteria:

* Patient has relapsed/progressed or is refractory for multiple myeloma following 1 previous line of therapy
* Measurable secretory multiple myeloma: measurable disease for secretory multiple myeloma is defined by at least one of the following measurements: serum monoclonal protein greater than or equal to 1 g/dl (> 10 gm/l) [10g/l], urine M-protein of ≥200 mg/24 hours
* Patient has a Karnofsky performance status of ≥ 60
* Patient has a life expectancy estimated at screening of at least 6 months
* Patient fulfills defined pretreatment laboratory requirements at and within 14 days before baseline

Exclusion Criteria:

* Patient received more than 1 previous line of therapy for multiple myeloma
* Patient has known allergy or hypersensitivity to bortezomib, Dexamethasone and/or Cyclophosphamide and/or Lenalidomide or any of the constituent compounds such as boron, mannitol, or lactose
* Patient has oligosecretory or non-secretory multiple myeloma
* Patient received nitrosoureas or any other chemotherapy (including thalidomide), clarithromycin, interferon within 6 weeks before enrolment. Note: subjects can have received thalidomide or interferon as maintenance therapy, according to local standard of care
* Patient received corticosteroids (> 10 mg/day prednisone or equivalent) within 3 weeks before enrolment. Note: subjects can have received steroids (dexamethasone or equivalent) as maintenance therapy according to local standard of care. In addition, subjects can have received a cumulative dose of up to 160 mg of dexamethasone or equivalent as emergency therapy within 3 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2008-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (42):
- France (4):
  - Bordeaux
  - Le Mans
  - Lille
  - Tours
- Germany (8):
  - Duisburg
  - Essen
  - Frankfurt (Oder)
  - Leipzig
  - München
  - Mÿnchen
  - Oldenburg
  - Ulm
- Greece (2):
  - Athens
  - Pátrai
- Hungary (5):
  - Budapest
  - Debrecen
  - Miskolc
  - Nyíregyháza
  - Szeged
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius Lt
- Poland (6):
  - Bialystok
  - Katowice
  - Krakow
  - Lodz
  - Warsaw
  - Wroclaw
- Serbia (4):
  - Belgrade
  - Kamenitz
  - Niš
  - Novi Sad
- Spain (4):
  - Barcelona
  - Madrid
  - Toledo
  - Valencia
- Turkey (Türkiye) (3):
  - Ankara
  - Istanbul
  - Izmir
- United Kingdom (3):
  - Bath
  - Edinburgh
  - London

REFERENCES:
- [Derived] Dimopoulos MA, Orlowski RZ, Facon T, Sonneveld P, Anderson KC, Beksac M, Benboubker L, Roddie H, Potamianou A, Couturier C, Feng H, Ataman O, van de Velde H, Richardson PG. Retrospective matched-pairs analysis of bortezomib plus dexamethasone versus bortezomib monotherapy in relapsed multiple myeloma. Haematologica. 2015 Jan;100(1):100-6. doi: 10.3324/haematol.2014.112037. Epub 2014 Sep 26. PMID 25261096

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 190 patients screened, 163 enrolled and received Bortezomib-Dexamethasone (VD) . Participants that completed cycles 1 to 4 were assessed for Response. Complete or Partial Responders were not randomized and continued on VD for cycles 5-8. Participants with Stable Disease (SD) were randomized to either VD, VDC, or VDR for cycles 5-8.
Groups:
- Cycle 1 to 4: Bortezomib + Dexamethasone (VD): bortezomib 1.3 mg/m2 IV bolus on Day 1, 4, 8, 11 in combination with dexamethasone 20 mg orally daily, on Days 1, 2, 4, 5, 8, 9, 11, 12 for 4 cycles
- Stable Disease: Bortezomib + Dexamethasone (VD): Stable disease after 4 cycles bortezomib + dexamethasone: bortezomib 1.3 mg/m2 IV bolus on Day 1, 4, 8, 11 in combination with dexamethasone 20 mg orally daily, on Days 1, 2, 4, 5, 8, 9, 11, 12 for cycle 5 to 8
- SD: Bortezomib+Dexamethasone+Cyclophosphamide (VDC): Stable disease after 4 cycles bortezomib + dexamethasone: bortezomib 1.3 mg/m2 IV bolus on Day 1, 4, 8 and 11 in combination with dexamethasone 20 mg orally daily, on Days 1, 2, 4, 5, 8, 9, 11, 12 and cyclophosphamide 500 mg, orally daily, days 1, 8 and 15 for cycle 5 to 8
- SD: Bortezomib+Dexamethasone+Lenalidomide (VDR): Stable disease after 4 cycles bortezomib + dexamethasone: bortezomib 1.3 mg/m2 IV bolus on Day 1, 4, 8 and 11 in combination with dexamethasone 20 mg orally daily, on Days 1, 2, 4, 5, 8, 9, 11, 12 and lenalidomide 10 mg orally daily from day 1 to day 14 for cycle 5 to 8
Period: Cycle 1 to 4
Arm/Group | Cycle 1 to 4: Bortezomib + Dexamethasone (VD) | Stable Disease: Bortezomib + Dexamethasone (VD) | SD: Bortezomib+Dexamethasone+Cyclophosphamide (VDC) | SD: Bortezomib+Dexamethasone+Lenalidomide (VDR)
Started | 163 (All participants started VD treatment for 4 cycles prior to local site response assessments) | 0 | 0 | 0
Completed | 135 (Of those completed, 120 subjects were assessed for response, 117 w/ Response or SD continued.) | 0 | 0 | 0
Not Completed | 28 | 0 | 0 | 0
Not completed — Death | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 0
Not completed — Progressive Disease | 6 | 0 | 0 | 0
Not completed — Adverse Event | 12 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0
Period: Randomization (Cycle 5) to Cycle 8
Arm/Group | Cycle 1 to 4: Bortezomib + Dexamethasone (VD) | Stable Disease: Bortezomib + Dexamethasone (VD) | SD: Bortezomib+Dexamethasone+Cyclophosphamide (VDC) | SD: Bortezomib+Dexamethasone+Lenalidomide (VDR)
Started | 98 (Responding patients (not randomized) who received 4 more cycles of VD) | 7 | 8 | 4
Completed | 63 | 4 | 7 | 4
Not Completed | 35 | 3 | 1 | 0
Not completed — Complete Response/Partial Response | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 5 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 1 | 0
Not completed — Adverse Event | 17 | 2 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0
Not completed — Other | 3 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: modified Intent to Treat Population consisting of all 163 participants with at least 1 dose and 1 post baseline efficacy assessment.: Complete and Partial Responders (non-randomized), n=144. Stable Disease (randomized to VD, VDC, and VDL), n=19.
Groups:
- All Study Participants: bortezomib 1.3 mg/m2 IV bolus on Day 1, 4, 8, 11 in combination with dexamethasone 20 mg orally daily, on Days 1, 2, 4, 5, 8, 9, 11, 12 for 4 cycles
Arm/Group | All Study Participants
Number analyzed (Participants) | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 86
Region of Enrollment [Number; unit: participants]
  France | 20
  Germany | 15
  Greece | 23
  Hungary | 2
  Lithuania | 9
  Poland | 19
  Serbia | 15
  Spain | 20
  Turkey | 19
  United Kingdom | 21

OUTCOME MEASURES:

1. Primary Outcome: Overall Best Confirmed Response
Description: Overall Best Confirmed Response is the best Overall Response Rate with borezomib-dexamathasone (+/-cyclophosphamide or lenalidomide) recorded between baseline and end of treatment. Response was assessed using the International Myeloma working Group (IMWG) Uniform Response Criteria and validated by an Independent Monitoring Committee.
Time Frame: Prior to treatment at day 1 of each cycle and at the end of treatment (day 21 of cycle 8), up to 168 days
Population: mITT: All patients with at least 1 dose and 1 post baseline assessment. Low powered study because necessary sample size for the randomized part could not be reached. Thus, data were analyzed and reported by combining the randomized groups with SD, (n=19). Data are missing for 21 patients in the non-randomized CR/PR group, n=123.
Measure: Number; unit: number of participants
Groups:
- Complete to Partial Response: Bortezomib + Dexamethasone: Complete, very good partial or partial response after 4 cycles bortezomib + dexamethasone: bortezomib 1.3 mg/m2 IV bolus on Day 1, 4, 8, 11 in combination with dexamethasone 20 mg orally daily, on Days 1, 2, 4, 5, 8, 9, 11, 12 for cycle 5 to 8
- Stable Disease After 4 Cycles: VD, VDC, VDL: Patients were treated with bortezomib 1.3 mg/m2 IV bolus on day 1, 4, 8 and 11 in combination with dexamethasone 20 mg orally on days 1, 2, 4, 5, 8, 9, 11, 12 for cycle 1 to 4. Patients with stable disease after these 4 cycles, were randomized at the start of cycle 5 and received either bortezomib 1.3 mg/m2 IV bolus on day 1, 4, 8 and 11 in combination with dexamethasone 20 mg orally, on days 1, 2, 4, 5, 8, 9, 11, 12 alone or in combination with cyclophosphamide 500 mg orally on days 1, 8 and 15 or lenalidomide 10 mg orally daily from day 1 to day 14 for cycle 5 to 8
Arm/Group | Complete to Partial Response: Bortezomib + Dexamethasone | Stable Disease After 4 Cycles: VD, VDC, VDL
Number analyzed (Participants) | 123 | 19
number of participants | 101 | 6

2. Secondary Outcome: Median Time to First Confirmed Response
Description: Time from start of treatment to the date of the first documentation of a confirmed response. Estimated using the Kaplan-Meier method. Response was assessed using the International Myeloma Working Group (IMWG) Uniform Response Criteria and validated by an Independent Monitoring Committee.
Time Frame: At Day 1 of each treatment cycle, at the End of Treatment visit until there is evidence of Progressive Disease or relapse from Complete Response (CR), up to 168 days
Population: mITT: All patients with at least 1 dose and 1 post baseline assessment. The non- randomized CR/PR group, n=144 for Time to First confirmed Response. Low powered study because necessary sample size for the randomized part could not be reached. Thus, data were analyzed and reported by combining the randomized groups with SD, (n=19).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Complete to Partial Response: Bortezomib + Dexamethasone | Stable Disease After 4 Cycles: VD, VDC, VDL
Number analyzed (Participants) | 144 | 19
days | 43.0 [43.0 to 58.0] | NA [152.0 to NA] — It is not possible to estimate the median time to first response or upper limit for the CI. This is because of the 19 subjects only 6 have an event, the majority is censored.

3. Secondary Outcome: Progression Free Survival
Description: Time from start of treatment to date of disease progression, relapse from CR or death. Estimated using the kaplan-meier method. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions", or similar definition as accurate and appropriate.
Time Frame: At Day 1 of each treatment cycle, at the End of Treatment visit until there is evidence of Progressive Disease or relapse from Complete Response (CR). Median Follow-Up of 16.9 months
Population: mITT: All patients with at least 1 dose and 1 post baseline assessment. The non-randomized CR/PR group, n=144. Low powered study because necessary sample size for the randomized part could not be reached. Thus, data were analyzed and reported by combining the randomized groups with SD, (n=19).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Complete to Partial Response: Bortezomib + Dexamethasone | Stable Disease After 4 Cycles: VD, VDC, VDL
Number analyzed (Participants) | 144 | 19
days | 311.0 [224.0 to 424.0] | 214.0 [198.0 to 234.0]

4. Secondary Outcome: Time to Progression
Description: Is calculated as the time from start of treatment to the date of the first observation of disease progression or relapse from CR. Deaths owing to causes other than progression not counted, but censored. Subjects who withdraw from the study or die will be censored at the time of last disease assessment. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0).
Time Frame: At Day 1 of each treatment cycle, at the End of Treatment visit until there is evidence of Progressive Disease or relapse from Complete Response (CR), Median Follow-up of 16.9 months
Population: mITT: All patients with at least 1 dose and 1 post baseline assessment. The non-randomized CR/PR group, n=144 for Time to First confirmed Response. Low powered study because necessary sample size for the randomized part could not be reached. Thus, data were analyzed and reported by combining the randomized groups with SD, (n=19).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Complete to Partial Response: Bortezomib + Dexamethasone | Stable Disease After 4 Cycles: VD, VDC, VDL
Number analyzed (Participants) | 144 | 19
days | 366.0 [281.0 to 475.0] | 214.0 [198.0 to 234.0]

5. Secondary Outcome: One Year Survival
Description: Percent Probability of Survival at 1 year from the start of treatment, estimated using Kaplan-Meier analysis.
Time Frame: At each visit from baseline to end of treatment. After treatment, monthly visit until progression or relapse or until the start of alternative MMY therapy, up to 1 year
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Complete to Partial Response: Bortezomib + Dexamethasone | Stable Disease After 4 Cycles: VD, VDC, VDL
Number analyzed (Participants) | 144 | 19
percent probability | 80 [73 to 87] | 89 [62 to 97]

6. Secondary Outcome: Overall Survival
Description: Is defined as the time interval from start of treatment to the date of death due to any cause. In the absence of confirmation of death (including subjects lost to follow-up), survival time will be censored at the last date the subject is known to be alive
Time Frame: At each visit from baseline to end of treatment. After treatment, monthly visit until progression or relapse or until the start of alternative MMY therapy. Further follow up by monthly phone call until the last patient was treated and followed for 1 year
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Complete to Partial Response: Bortezomib + Dexamethasone | Stable Disease After 4 Cycles: VD, VDC, VDL
Number analyzed (Participants) | 144 | 19
days | NA [888.0 to NA] — this value could not be calculated due to the limited number of events | NA [982.0 to NA] — this value could not be calculated due to the limited number of events

ADVERSE EVENTS:
Time Frame: From signing of informed consent until 30 days after the last dose of study medication (approximately 7 months) or longer if considered related to study medication.
Description: Due to the high response rate of the bortezomib-dexmathasone (VD) in the first four cycles, not enough patients could be randomized to the sequential therapies in cycles 5-8 to allow us to evaluate safety data according randomization or intervention. Thus, adverse events were analyzed by combining (randomized) participants with SD After 4 Cycles.
Arm/Group | Complete to Partial Response: Bortezomib + Dexamethasone | Stable Disease After 4 Cycles: VD, VDC, VDL
Serious Adverse Events (participants affected / at risk) | 59/144 | 6/19
Other Adverse Events (participants affected / at risk) | 137/144 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Complete to Partial Response: Bortezomib + Dexamethasone (N=144) | Stable Disease After 4 Cycles: VD, VDC, VDL (N=19)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 2 (3) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic Stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial Rupture (Vascular disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Shock Haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (7) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Cardiac Failure (Cardiac disorders) | 3 (3) | 1 (3)
Myocardial Infarction (Cardiac disorders) | 3 (3) | 0 (0)
Atrial Fibrilation (Cardiac disorders) | 3 (3) | 0 (0)
Agina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis Ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Oedema Peripheral (General disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 9 (10) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 3 (3) | 1 (1)
Bronchitis (Infections and infestations) | 3 (4) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Subcutaneous Abscess (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Rotavirus (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar Abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumomonia Pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0)
Cervical Vertebral Fraction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Liver Function Test Abnormal (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebellar Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient Ischemic Attack (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Chest Wall Abscess (Infections and infestations) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Complete to Partial Response: Bortezomib + Dexamethasone (N=144) | Stable Disease After 4 Cycles: VD, VDC, VDL (N=19)
Thrombocytopenia (Blood and lymphatic system disorders) | 52 (216) | 8 (22)
Anaemia (Blood and lymphatic system disorders) | 29 (79) | 6 (14)
Neutropenia (Blood and lymphatic system disorders) | 10 (20) | 2 (7)
Leukopenia (Blood and lymphatic system disorders) | 8 (37) | 1 (1)
Conjunctivitis (Eye disorders) | 8 (10) | 2 (3)
Constipation (Gastrointestinal disorders) | 45 (81) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 45 (66) | 5 (5)
Nausea (Gastrointestinal disorders) | 16 (23) | 3 (5)
Abdominal Pain (Gastrointestinal disorders) | 8 (8) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 11 (15) | 1 (2)
Vomiting (Gastrointestinal disorders) | 10 (11) | 1 (1)
Oedema Peripheral (General disorders) | 38 (49) | 5 (11)
Fatigue (General disorders) | 37 (62) | 0 (0)
Asthenia (General disorders) | 29 (36) | 4 (5)
Pyrexia (General disorders) | 15 (15) | 4 (12)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 13 (17) | 3 (3)
Herpes Zoster (Infections and infestations) | 12 (12) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 12 (17) | 2 (2)
Nasopharyngitis (Infections and infestations) | 9 (11) | 1 (1)
Oral Candidiasis (Infections and infestations) | 8 (10) | 2 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (11) | 3 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 21 (28) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (15) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 11 (19) | 1 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 14 (25) | 2 (3)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 11 (13) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 29 (80) | 4 (11)
Polyneuropathy (Nervous system disorders) | 26 (40) | 2 (5)
Neuralgia (Nervous system disorders) | 22 (33) | 4 (6)
Neuropathy Peripheral (Nervous system disorders) | 21 (42) | 0 (0)
Paraesthesia (Nervous system disorders) | 19 (27) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 13 (19) | 2 (3)
Dizziness (Nervous system disorders) | 13 (17) | 1 (2)
Headache (Nervous system disorders) | 9 (13) | 0 (0)
Insomnia (Psychiatric disorders) | 15 (19) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (27) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 3 (4)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 1 (1)
Hypotension (Vascular disorders) | 11 (17) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 9 (15) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 8 (11) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (3)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 1 (1)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5) | 1 (3)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Cellulitis (Infections and infestations) | 3 (6) | 1 (1)
Oral herpes (Infections and infestations) | 3 (3) | 1 (1)
Oral infection (Infections and infestations) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 3 (3) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (6) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 6 (8) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 2 (3) | 1 (1)
Confusional state (Psychiatric disorders) | 5 (5) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 2 (3) | 2 (2)
Haematoma (Vascular disorders) | 1 (1) | 1 (1)
Aortic elongation (Vascular disorders) | 0 (0) | 1 (1)
Trigeminal Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
The response rate of bortezomib in combination with dexamethasone after 4 cycles was much higher than originally assumed. Therefore the sample size of the randomized groups is too small for further statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days